CLINICAL TRIAL: NCT05132686
Title: Effects of Intermittent Energy Restriction on Intra-Abdominal Fat and the Gut Microbiome: A Randomized Trial
Brief Title: The Healthy Diet and Lifestyle Study II
Acronym: (HDLS2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Hawaii Cancer Research Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LEMARCHAND-2021-2; 1R01CA258179-01A1 (NIH)
Record Dates: First submitted 2021-09-20; First posted 2021-11-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Intra-Abdominal Fat
Keywords: Visceral Adipose Tissue, Visceral Fat; Intermittent energy restriction; Randomized Controlled Trial; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail. Participants will be randomized to either intermittent energy restriction (IER) and Mediterranean diet (MED) / IER+MED or the daily energy restriction (DER) and the Mediterranean diet / (MED/DER).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be provided with healthful dietary information but will not be told what diets their diet plans are based on. Participants in the IER+MED diet group will be told they are on diet plan 1 and participants in the MED/DER diet group will be told they are on diet plan A. The dietitians will know which diet plan each participant is on, however; all other clinic staff who assess outcome measures will be blinded to each participant's diet group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent energy restriction (IER) + Mediterranean diet (MED) or IER+MED (Experimental): The IER+MED group intervention will be to restrict 70% energy (25%, 45% and 30% distribution of protein, carbohydrate, and fat, respectively) on 2 days and follow a MED diet (25%, 45%, 30%) and meet their estimated energy requirement (EER) for the other 5 days each week. This would be equivalent to an over-all 20% daily energy restriction. Participants will also be asked to follow a moderate exercise program (1 hour of walking five days a week).
  Interventions: Behavioral: IER+MED
- Mediterranean diet (MED) + daily energy restriction (DER) or MED/DER (Experimental): The MED/DER group intervention will restrict 20% energy (25%, 45% and 30% distribution of protein, carbohydrate, and fat, respectively) continuously. Participants will also be asked to follow a moderate exercise program (1 hour of walking five days a week).
  Interventions: Behavioral: MED/DER

INTERVENTIONS:
Behavioral: IER+MED — Over a 6 month period follow a euenergetic Mediterranean diet 5 days per week and a 20% energy restriction over 2 contiguous days as a 70% energy restriction using the same macronutrient distribution of 45% carbohydrate, 25% energy from protein, and 30% energy from fat. For each participant a tailored diet plan is created based on sex, weight, height, and age. Complete a 1 hour walk five days per week.
  Other Names: The Healthy Diet and Lifestyle Study II (HDLS2)
  Arms: Intermittent energy restriction (IER) + Mediterranean diet (MED) or IER+MED
Behavioral: MED/DER — Over a 6 month period follow a Mediterranean diet 7 days per week with a 20% energy restriction 7 days a week using the macronutrient distribution of 45% carbohydrate, 25% energy from protein, and 30% energy from fat. For each participant a tailored diet plan is created based on sex, weight, height, and age. Complete a 1 hour walk five days per week.
  Other Names: The Healthy Diet and Lifestyle Study II (HDLS2)
  Arms: Mediterranean diet (MED) + daily energy restriction (DER) or MED/DER

SUMMARY:
Intermittent energy restriction (IER) may have important advantages over daily energy restriction (DER) in producing sustained weight loss and reducing cancer risk. IER is already being promoted with limited evidence, thus, additional evidence is urgently needed from rigorously conducted clinical trials. IER has been proposed to invoke a greater metabolic shift to fat metabolism than DER and preferentially reduce central obesity. The Investigators adapted the IER and the Mediterranean diet (MED) approach which have been recommended as a healthy weight-loss diet in the management of non-alcoholic fatty liver disease, for an ethnically diverse population. The effectiveness was compared to an active comparator (DASH diet) in reducing overall and visceral adiposity in a randomized trial among 60 middle-aged adults with visceral obesity. This 12-week pilot demonstrated the feasibility and safety of IER and the culturally-adapted MED [NCT03639350]. The six-month randomized trial will demonstrate the superiority of IER over DER in reducing fat and total fat mass, and in improving cancer-related biomarkers and gut microbiome functions. This longer trial, to confirm safety and superiority of IER over DER in reducing VAT and liver fat will expand our understanding of adherence to IER and its effect on the gut microbiome as a possible mediator of systemic inflammation. The Investigators will conduct a 24-week randomized trial of IER+MED vs. MED/DER among 260 middle-aged adults of East-Asian, Native Hawaiian and other Pacific Islanders or White ethnicity with high VAT. The primary research question is whether a diet plan combining IER and the MED dietary pattern will be superior to MED/DER in reducing abdominal MRI-measured visceral and liver fat and dual-energy X-ray absorptiometry (DXA) measured total adiposity. The Healthy Diet and Lifestyle Study II (HDLS2) will recruit 312 men and women from the general population with VAT at or above the population-median (men: ≥90 cm2; women ≥80 cm2) and randomize them to the IER+MED or MED/DER diet (156 per group). The IER+MED group will follow IER for two consecutive days (70% energy restriction) and total energy MED diet for the other five days of the week, reaching an overall 20% energy restriction. The MED/DER group will be prescribed a 20% daily energy restriction. With an expected attrition rate of ~16% (10% in Pilot), the investigators expect 130 participants per group to complete the study.

DETAILED DESCRIPTION:
Goal: This study proposes a 24-week randomized trial of intermittent energy restriction (IER) and the Mediterranean diet (MED), IER+MED, compared to daily energy restriction (MED/DER) among 260 middle-aged adults of East-Asian, Native Hawaiian and other Pacific Islanders or white ethnicity with high visceral fat (VAT) and liver fat.

1. To investigate whether a diet plan combining IER+MED will be superior to MED/DER in reducing abdominal visceral and liver fat and total adiposity among a multiethnic, at-risk, adult population. The Healthy Diet and Lifestyle Study II (HDLS2) plans to recruit 312 men and women from the general population with VAT at or above the population-median (men: ≥90 cm2; women ≥80 cm2) and randomize them to the IER+MED or MED/DER diet (156 per group). The IER+MED group will follow IER for two consecutive days (70% energy restriction) and a total energy MED diet for the other five days of the week, reaching an overall 20% energy restriction. The MED/DER group will be prescribed a 20% daily energy restriction. The expected attrition rate is ~16%, thus 130 participants per group are expected to complete the study.
2. To determine if the IER+MED compared to the MED/DER influences intermediate markers: cancer-related blood biomarkers and the gut microbial community structure and function.
3. To assess behavioral predictors of adherence to the prescribed IER+MED and DER/MED. To test modifications to psychosocial constructs being associated with adherence differently between IER+MED and MED/DER.

Design: The HDLS2 is a parallel, randomized, trial to compare the effects of two diets over 24-weeks: the IER+MED diet pattern vs. the MED/DER daily energy restriction diet pattern. For randomization, biostatisticians will prepare a blocked randomization schedule, stratified by men/women, the three ethnic groups, age <50 and 50+ y for men, menopausal status for women (based on any periods in the last 12 months), and two VAT groups (high, 80-150 cm2 or very high, ≥150 cm2). The randomization procedure will be conducted using opaque, sealed, sequentially numbered envelopes each containing assignment with equal probability to one of the two dietary interventions. The participants and measurement staff will be masked from the moniker of the assigned dietary intervention. The dietitians will coordinate and conduct the intervention activities using four face to face meetings (or an alterative if needed), and 12 remote meetings using phones or communication platforms (eg. Zoom). Every effort will be made for each participant to stay with the same dietitian. Enrollment of 156/study arm and completion of the intervention activities will take place over 3.5 years.

The research will be carried out in the University of Hawaii Cancer Center (UHCC) Translational Research Clinic, Nutrition Education Center, and Metabolic Kitchen, as well as the University of Hawaii (UH) Magnetic Resonance Imaging (MRI) Research Center. Each of these units have approved common guidelines addressing specific guidance for the coronavirus disease (COVID-19) screening of staff and research participants prior to the visit, upon arrival to the clinic, entry to the clinic, and post appointment guidelines.

Recruitment, clinic, and imaging staff will be blinded to randomization and intervention activities. Likewise, other than baseline demographic information, the intervention staff (dietitians) will be blinded to assessment measures of the study participants (with the exception of body weight, which is needed for the dietary prescriptions). Volunteers will be recruited among Oahu residents using advertising, media exposure, community and workplace presentations, and referrals from clinical partners. Main eligibility criteria were informed by the pilot study. Assuming a ~16% drop-out rate to yield 260 participants completing the 6-month intervention. The first recruits will start in October 2021, with the goal of recruiting 16 participants/month (except mid Nov through first week of Jan).

Assessing dietary intervention adherence: To assess dietary intervention adherence, dietary intake of energy, fat (monounsaturated fat (MUFA), polyunsaturated fat (PUFA) and saturated fat (SAT)), carbohydrate, protein, dietary fiber and alcohol will be assessed prior to the first week of intervention, then every month thereafter. The participants will complete their 4-day mobile Food Record (mFR) the week before the clinic visits at Week 12 (midpoint), Week 24 (end of intervention) and Week 48 (maintenance). This allows the dietitians to proceed with efficient participant sessions. The images captured using the mFR app include before and after images of each eating occasion, time, location, and other contextual information. Some foods are difficult to distinguish in images; therefore, a questionnaire at the first visit addressing type of oils, milk, and other salient foods will be administered. Data collected with the mFR app facilitates translation to better address eating behaviors and assess effectiveness of interventions. The Investigators expect that most participants will have a smart phone and will be able to download the app; however, the Investigators will loan devices if needed. For the MED/DER group, the average intakes will be computed across the 4 days. For the IER+MED, the intakes will be computed separately for the 2 IER days and for the 2 MED days, as well as by overall means weighting IER means by 2/7 and the MED means by 5/7. The percentage of the recommended amount for energy and the macronutrients will be computed for each week, and averaged across weeks. Similarly, changes in physical activity over time, in particular the average minutes of moderate/vigorous activity, based on the physical activity questionnaire and accelerometer data, will be examined across baseline, 4 weeks, 12 weeks, and 24 weeks.

Advice, support and monitoring in both diet groups: The 16 dietary and physical activity counseling sessions will be completed by the dietitians with each participant. Foods eaten as part of the IER+MED and MED/DER diets will be self-selected by the participants. Both groups will receive clear instructions on how to follow their allocated diet in a face-to-face dietary consultation or remotely with one of the research dietitians (45-60 minutes). Both arms will also receive comprehensive written instructions on how to follow the diets at home, including recommended portion sizes and recipes and suggested meal plans. Both groups will receive appropriate behavioral techniques to promote adherence to diets. For non-clinic visits, participants in both groups will be contacted using the participants preferred method of contact, e.g, phone, communication platform (eg. Zoom), with their allocated dietitian one week after randomization to check they have started the diet, to assess their understanding of the diet and to provide any troubleshooting advice. Throughout the trial, all participants will be advised to become more active and will receive information providing a program of walking at least one hour five days per week. The IER+MED group will be encouraged to walk on the non-IER days. All will be advised and shown how to do resistance exercise as bicep curls and upper-body resistance exercises (i.e., seated leg press and overhead press using a provided resistance band). The recommendation is 2 nonconsecutive days per week as 3 sets of 8-10 repetitions. Cooking demonstration classes using the metabolic kitchen in the UHCC which has an adjoining Nutrition Education space with overhead cameras to complement the view of the activities in the kitchen will be conducted. After enrollment of the first group of participants, classes will be offered every month to accommodate each study arm separately, with content aligned with the assigned dietary pattern.

Statistical Considerations. Statistical analysis will be conducted with the Epidemiology Program, UHCC. The data management system developed for the Pilot HDLS will be adapted to monitor recruitment, study milestones, specimen collection, inventory, and data entry systems. For this aim, the Investigators will compare the changes in adiposity outcomes over the 24-week intervention between the two intervention groups using an intention-to-treat approach. In particular, the following outcomes will be considered: Primary: MRI VAT, percent liver fat; Secondary: body weight, BMI, DXA total body fat, percentage body fat, total DXA muscle mass, trunk fat, SAT area, percent pancreatic fat, fat free mass (FFM), VAT/SAT ratio, and DXA VAT. A linear mixed model will be fit for each outcome with fixed independent variables of intervention arm, time (baseline, Weeks 12, 24), interaction terms between group and time, and any adjustment variables needed to account for imbalance in participant characteristics between groups and a random effect for participant. Covariate-adjusted means and 95% confidence intervals will be computed for each arm and time point. Effect size will be computed as the difference between the two intervention arms in change in the means at Week 12 and at Week 24 from baseline. The primary test of the intervention effect will be based on differences in means at Week 24 using a Wald test of the interaction terms at this time point. While the Investigators will strive to minimize withdrawals and missing data, the investigators will also investigate whether missing data have biased the results.

Post-Study: At the end of the study all participants will be offered advice on continued weight loss and/or weight loss maintenance if they have reached a target weight and this is appropriate. This will include advice regarding their preferred diet, i.e. IER+MED or MED/DER.

Ethical Considerations: The study will be preformed in accordance with the ethical principles in the Declaration of Helsinki and the University of Hawaii operational and ethical guidelines for research and other applicable regulatory requirements.

Participant information and consent: Consent to enter the study will be sought from each participant only after a full explanation has been given, information has been provided and time allowed for consideration. The right of the participant to refuse to participate without giving reasons will be respected.

Discontinuation and withdrawal: Participants are free to withdraw from the study at any time, without prejudice to further treatment. Participants may also be discontinued from the study at any time, at the discretion of the investigator. Requests by the participant to be withdrawn for the study should be made through the principal investigator.

Confidentiality: After the participant has consented, any information from the study will be stored on a secure password-protected server that will be accessible only to the research team. Trial data on anthropometry and activity data will be kept on a secure server at the UHCC. The food & beverage images from the 4-day mobile food records with be kept on a secure server.

Data Handling and Record Keeping. All data will be kept strictly confidential. Any individual volunteering to participant will be assigned a code number, with the link to identifying information only available to the few study staff that require this information. Identifying information will be maintained in separate secure computer files from the remainder of the data. All forms will be stored in locked file cabinets, and those with identifying information will be stored separately from the other forms. No analysis will ever identify participants individually.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-69 years old
* BMI between 25-40 kg/m2
* Currently non-smoking
* No serious health issues
* Fully vaccinated for COVID-19
* Normal blood chemistry profile
* East Asian (Chinese, Japanese, Korean), Filipino, Native Hawaiian/other Pacific Islander or white/European ancestry
* Non-drinkers / low habitual drinkers, i.e., men ≤15 drinks per week, women ≤10 drinks per week
* Volunteers living on the island of Oahu
* For peri-menopausal women, the investigators will require that they had their last period at least 1 year before baseline)
* DXA VAT ≥90 cm2 for men and ≥80 cm2 for women
* Able to read, speak, and write in English

Exclusion Criteria:

* Pregnancy
* Contraindication to MR imaging (e.g. pacemaker, claustrophobia, metal implants)
* Previous surgery to remove any part of the small intestine, colon or rectum (e.g.

ileostomy or colectomy) or an amputation of a leg or arm.

* For women, taking any anti-estrogen medications (e.g tamoxifen, Nolvadex, Istubal, Valodex)
* For men, taking any anti-androgen medications (e.g., Eulexin (flutamide); Anandron or Nilandron (nilutamide); Casodex (bicalutamide); Proscar or Propecia (finasteride); Avodart (dutasteride); or bexlosteride, izonsteride, turosteride, episteride).
* Diagnosis of Type 1 diabetes or Type 2 diabetes and taking insulin for treatment
* Diagnosis of thyroid conditions under treatment with hormones or medications.
* Serious health issues such as dialysis, organ transplant, celiac disease, Crohn's disease, chronic liver disease, active case of hepatitis B or C, chronic kidney disease, or any condition that, in the opinion of the investigator, is a contraindication to participation.
* Previous problem with fasting blood collection
* Cannot exercise (walk) for up to 1hr/day

Deferral Criteria :

Volunteers with the following conditions will be called back after the specified duration:

* Treatments in past 6 months: chemotherapy or radiation of abdomen/pelvis; corticosteroid hormones; prescription weight loss drugs; estrogen/androgen receptor blockers
* Substantial weight change (>20lbs) in past 6 months
* Antibiotic use in past 3 months
* Colonoscopy, sigmoidoscopy, colon irrigation/bowel cleaning in the past 3 months
* MRI/CAT scan with contrast in the past 2 weeks

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Abdominal magnetic resonance imaging (MRI) to measure visceral fat and liver fat | Week 24
  To investigate whether a diet plan combining intermittent energy restriction (IER) and a Mediterranean diet (MED) dietary pattern (IER+MED) will be superior to a MED diet and daily energy restriction (DER) (MED/DER) in reducing abdominal MRI-measured visceral and liver fat.
Dual-energy X-ray absorptiometry (DXA) scan for total adiposity | Week 24
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing DXA-measured total adiposity.

SECONDARY OUTCOMES:
DXA scan for total adiposity at week 48 (24 weeks post trial) | Week 48
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing long term DXA-measured total adiposity, after 24 weeks post clinical trial.
Measured body weight at end of trial | Week 24
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing body weight at the end of the trial.
Measured body weight at week 48 (24 weeks post trial). | Week 48
  To investigate whether the diet plan IER+MED will be superior to MED/DER in maintaining long term body weight loss after 24 weeks post clinical trial.
Computed body mass index (BMI) at end of trial. | Week 24
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing body weight at the end of the trial.
Computed body mass index (BMI) (24 weeks post trial) | Week 48
  To investigate whether the diet plan IER+MED will be superior to MED/DER in maintaining long term body weight loss after 24 weeks post clinical trial.
Measured waist- and hip-circumferences at end of trial. | Week 24
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing body circumference measures associated with visceral adiposity at the end of trial.
Measured waist- and hip-circumferences (24 weeks post trial) | Week 48
  To investigate whether the diet plan IER+MED will be superior to MED/DER in maintaining long term body weight loss after 24 weeks post clinical trial.
Fat mass, computation of fat mass using completed measurement values at end of trial. | Week 24
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing fat mass associated with visceral adiposity at the end of trial.
Fat mass, computation of fat mass using completed measurement values (24 weeks post trial) | Week 48
  To investigate whether the diet plan IER+MED will be superior to MED/DER in reducing fat mass associated with visceral adiposity at the end of trial in maintaining long term body weight loss after 24 weeks post clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Loic Le Marchand, MD, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will consist of cleaned, anonymized, and analyzable datasets. Data will be made available to secondary researchers. Specific data to be shared will be de-identified addressing secondary intervention topics. Data sharing will become available after publication of the three primary results and then will be available indefinitely. Data will be shared with investigators when proposed research has received Institutional Review Board (IRB) approval. Also, to be provided, study protocol, original statistical analysis plan, informed consent form, clinical study reports, and others will be considered as needed. Qualified researchers with IRB approval would be eligible to receive the data. Include at least one original member of the HDLS2 as a co-author. The Investigators will share experimental and behavioral data associated with the study participants by depositing these data with the University of Hawaii Biostatistics Shared Resource.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting information will become available at least 2 years after the study ends and the 3 designated papers are submitted.
Access Criteria: Qualified researchers who have received IRB approval would be eligible to receive data.
  At least one original member of the Healthy Diet and Life Style Study HDLS2 would need to be included as a co-author.
  The Investigators will share experimental and behavioral data associated with the study participants by depositing these data with the University of Hawaii Biostatistics Shared Resource.
  To prepare the materials, the usual fees will be implemented. Information can be accessed at: The University of Hawaii Cancer Center, Biostatistics Shared Resource.
URL: http://uhcancercenter.org/research/shared-resources/biostatistics

REFERENCES:
- [Result] O'Reilly H, Panizza CE, Lim U, Yonemori KM, Wilkens LR, Shvetsov YB, Harvie MN, Shepherd J, Zhu FM, Le Marchand L, Boushey CJ, Cassel KD. Utility of self-rated adherence for monitoring dietary and physical activity compliance and assessment of participant feedback of the Healthy Diet and Lifestyle Study pilot. Pilot Feasibility Stud. 2021 Feb 11;7(1):48. doi: 10.1186/s40814-021-00786-3. PMID 33573693
- [Result] Panizza CE, Wong MC, Kelly N, Liu YE, Shvetsov YB, Lowe DA, Weiss EJ, Heymsfield SB, Kennedy S, Boushey CJ, Maskarinec G, Shepherd JA. Diet Quality and Visceral Adiposity among a Multiethnic Population of Young, Middle, and Older Aged Adults. Curr Dev Nutr. 2020 May 26;4(6):nzaa090. doi: 10.1093/cdn/nzaa090. eCollection 2020 Jun. PMID 33959689
- [Derived] Lewis MY, Yonemori K, Ross A, Wilkens LR, Shepherd J, Cassel K, Stenger A, Rettenmeier C, Lim U, Boushey C, Le Marchand L. Effect of Intermittent vs. Continuous Energy Restriction on Visceral Fat: Protocol for The Healthy Diet and Lifestyle Study 2 (HDLS2). Nutrients. 2024 May 14;16(10):1478. doi: 10.3390/nu16101478. PMID 38794715